CLINICAL TRIAL: NCT05526937
Title: The Effect of Sprouting of Wheat on Postprandial Glycemic and Satiety Responses of Wheat Bread Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 22-06-26
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Blood Sugar
MeSH Terms: interventions — Bread

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sprouted wholemeal bread (Experimental)
  Interventions: Other: Bread
- Unsprouted wholemeal bread (Active Comparator)
  Interventions: Other: Bread
- White bread (Placebo Comparator)
  Interventions: Other: Bread

INTERVENTIONS:
Other: Bread — Bread portions of 50 gram available carbohydrates.

SUMMARY:
The objective of this study is to investigate the effect of inclusion of 50% sprouted wheat wholemeal in a bread recipe on the postprandial glycemic and satiety responses, as well as on appetite-related sensations and acceptability of the developed products relative to a product made with a similar unsprouted wheat recipe.

DETAILED DESCRIPTION:
This study is a randomized crossover trial involving three different bread products. At each study visit, capillary blood glucose will be measured at fasting, and then 15, 30, 45, 60, 90, and 120 minutes following the start of ingestion of the study food. Visual analogue scales will be used to assess appetite and fullness sensations at fasting, and then 30, 60, 90 and 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age 18-40 years
* Normal non-fasting plasma glucose (<7.9 mmol/L but not below 3.3 mmol/L)
* BMI ranging from 18.5 to 27.9 kg/m2
* Regular consumer of wheat-based bread products (>1x per week).

Exclusion Criteria:

* Smoking or regular use of recreational drugs (marijuana, ecstasy, LSD, magic mushrooms etc.)
* Heavy alcohol use (defined as typically >14 drinks per week or >4 drinks on one occasion)
* Restrained eater (>16) as defined by the questionnaire at screening (Appendix E: Three Factor Eating Questionnaire, Stunkard et al.,1985)
* Unusual sleep patterns (Shift-worker, or sleeps 4 hours or less regularly) or irregular breakfast consumption.
* Recent (i.e. >4 kg in previous 3 months) or intended weight loss or gain
* Food allergies or any life-threatening allergy (food or otherwise)
* Gluten intolerance or sensitivity
* Medications known to affect glucose tolerance (excluding oral contraceptives)
* Presence of disease or drug(s) which influence digestion and absorption of nutrients; including steroids, protease inhibitors or antipsychotics.
* Inability to adhere to Study Protocols

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | 2 hours
  Capillary blood glucose

SECONDARY OUTCOMES:
Postprandial satiety response | 2 hours
  Hunger, Fullness, Desire to Eat and Prospective Food Consumption questions using Visual Analogue Scales (100 mm lines). Answers are measured and scored from 0 (not at all) to 100 (extreme).

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No